CLINICAL TRIAL: NCT00250861
Title: A Randomized Phase II Trial of Outpatient Immunotherapy With Rituximab and Aldesleukin (IL-2) vs. Rituximab Alone for CD20 Positive Aggressive Non-Hodgkin's Lymphoma Following High Dose Therapy With Autologous PBSC Rescue
Brief Title: Trial of Outpatient Immunotherapy With Rituximab and Aldesleukin (IL-2) vs. Rituximab Alone for Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment.
Sponsor: US Oncology Research (Industry)
Collaborators: Chiron Corporation (Industry); Fred Hutchinson Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US-I-IL2-04-029
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; aldesleukin

INTERVENTIONS:
Drug: Rituximab
Drug: Aldesleukin

SUMMARY:
The purpose of this research study is to find out if treatment with rituximab in combination with aldesleukin (compared to rituximab alone) decreases the risk of cancer returning, as well as determining what other effects (good and bad) this drug combination has on NHL. Rituximab and aldesleukin are not approved in combination by the Food and Drug Administration (FDA) for the treatment of non-Hodgkins lymphoma; however, Rituximab is approved for use by itself to treat NHL.

ELIGIBILITY:
INCLUSION CRITERIA:

A patient will be eligible for inclusion in this study if s/he meets all of the following criteria:

* Has previously undergone BEAC or BEAM autologus SCT with PBSC rescue for any stage aggressive B-cell NHL, including transformed indolent NHL or mantle cell lymphoma according to REAL classification - only B-cell lymphomas are permitted.
* ECOG performance status 0-1.
* Previously histological documented CD20 +NHL.
* Is greater than 18 years of age.
* Is 30-100 days from autologous peripheral blood stem cell transplant.
* Must meet laboratory values (see protocol for values): Absolute neutrophils, hemoglobin and platelets.
* Has a negative serum pregnancy test within 7 days prior to trial registration (only for female patients of childbearing potential).
* If fertile, patient (male or female) has agreed to use physician-approved method of birth control to avoid pregnancy for the duration of the study and for a period of 3 months thereafter.
* Has signed a Patient Informed Consent Form.
* Has signed a Patient Authorization Form (HIPAA).

EXCLUSION CRITERIA:

Patients will be taken off treatment if any of the following occur:

* ECOG PS >2.
* A history of hypersensitivity to study drugs, or any component thereof, or anaphylactic history to murine protein.
* Manifested cardiac complications during transplant, including arrthymias, congestive heart failure, angina, or myocardial infarct, or had a decreased LVEF to <45% prior to transplant
* On systemic corticosteroids.
* Diffusion capacity <60% (corrected) and has decreased 30% or more following transplant
* Documented disease progression (See Section 10.1.6 for definition).
* Active infection, and/or is known to be seropositive for hepatitis B, hepatitis C, or HIV
* Pericardial effusion, pleural effusions, or ascites.
* A history of very aggressive NHL, such as Burkitt's or atypical Burkitt's lymphoma
* Receiving concurrent immunotherapy or rituximab therapy.
* Previously received a solid organ transplant.
* History of CNS involvement.
* A serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
* A history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs.
* A pregnant or nursing woman.
* Unable to comply with requirements of study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2005-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Williams, MD, Principal Investigator — US Oncology Research
Locations (21):
- United States (21):
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Kansas City Cancer Centers-Central, Kansas City, Missouri
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Cancer Center, Arlington, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - San Antonio Tumor & Blood Clinic, Fredericksburg, Texas
  - Texas Oncology, PA, Garland, Texas
  - Longview Cancer Center, Longview, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Fairfax Northern VA Hem-Onc PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Pudget Sound Cancer Center-Seattle, Seattle, Washington
  - Cancer Care Northwest-North, Spokane, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington